CLINICAL TRIAL: NCT04801095
Title: A Phase I, Open-label, Multicenter, Dose-escalation and Dose-expansion Study to Investigate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Efficacy of WM-S1-030 in Patients With Advanced Solid Tumors
Brief Title: A Phase I Study of WM-S1-030 in Patients With Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wellmarker Bio (Industry)
Collaborators: Covance (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WMS1030-101
Record Dates: First submitted 2021-03-04; First posted 2021-03-16 (Actual); Last update posted 2022-09-16 (Actual); Status verified 2022-09

CONDITIONS: Advanced Solid Tumor; Metastatic Solid Tumor; Colorectal Cancer; Lung Cancer; Pancreatic Cancer; Cholangiocarcinoma; Head and Neck Cancer
MeSH Terms: conditions — Neoplasm Metastasis; Colorectal Neoplasms; Lung Neoplasms; Pancreatic Neoplasms; Cholangiocarcinoma; Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- WM-S1-030 (Experimental): Dose escalation (part 1) and Dose expansion (part 2)
  Interventions: Drug: WM-S1-030

INTERVENTIONS:
Drug: WM-S1-030 — WM-S1-030 orally administered once daily (QD) for 28 days of each cycle.

SUMMARY:
This study evaluates the safety, tolerability, pharmacokinetics, pharmacodynamics, and efficacy of WM-S1-030 in patients with advanced solid tumors.

DETAILED DESCRIPTION:
This is a Phase I, open-label, multicenter, dose-escalation, and dose-expansion study of WM-S1-030 in patients with advanced or metastatic solid tumors. The study will be conducted in 2 parts; a dose-escalation phase (Part 1) and a dose-expansion phase (Part 2). Part 1 will investigate oral administration of WM-S1-030 as monotherapy. Once the MTD or recommended dose is identified in Part 1, additional patients will be enrolled into Part 2 to further investigate efficacy, safety, PK, pharmacodynamics, dosing interval or schedule, and food effect on the single-dose PK of WM-S1-030.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥18 years.
2. Able and willing to sign the informed consent form (ICF).
3. Have at least 1 evaluable lesion based on Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.
4. Have histologically or cytologically confirmed locally advanced unresectable or metastatic solid tumor which has progressed after treatment with standard therapies and for which no effective standard therapy is available or patient has refused, has a contraindication, or is intolerant to standard therapies.
5. Have Eastern Cooperative Oncology Group (ECOG) performance status ≤2.
6. Must have archived frozen tissue available (collected within 3 months before screening) or consent to a pre-treatment biopsy.
7. Must be willing to consent to up to 2 on-treatment biopsies.
8. Have a life expectancy of at least 12 weeks.
9. Have adequate hematological functions and blood coagulation.
10. Have adequate hepatic function at screening.
11. Have adequate renal function at screening.
12. QT interval corrected for heart rate using Fridericia's method ≤470 msec.
13. Agree to abide by contraception requirements.
14. Body mass index between 18 and 35 kg/m2 (exclusive)

Exclusion Criteria:

1. Have received any prior approved or investigational treatment with RON and/or tyrosine-protein kinase Met (hepatocyte growth factor receptor) such as rilotumumab or crizotinib.
2. Have received any cytotoxic chemotherapy, investigational agent (or medical device), anticancer drug, hormone therapy, or radiation therapy for treatment within 4 weeks or therapeutic radiopharmaceuticals taken within 8 weeks prior to the first administration of IP. Point (or limited) radiation to a site of bone pain, with the exception of patients receiving radiation to more than 30% of the bone marrow, will be allowed.
3. Have known hypersensitivity to WM-S1-030 and/or excipient.
4. Have ≥ Grade 2 unresolved toxicity related to prior anticancer therapy excluding alopecia.
5. Have received drugs or herbal supplements within 2 weeks prior to the first administration of IP which are known to be inhibitors or inducers of cytochrome P450 (CYP)3A4 including, but not limited to, cannabinoids, ketoconazole, itraconazole, posaconazole, voriconazole, rifampicin, phenytoin, St. John's Wort, carbamazepine, or hyperforin.
6. Have any primary central nervous system (CNS) tumors or known CNS metastases unless clinically stable (defined as without evidence of progression by imaging at least 4 weeks prior to the first administration of IP; any neurologic symptoms have returned to baseline), no evidence of new or enlarging brain metastases, and not using steroids or seizure medications (unless on stable doses) for at least 7 days prior to the first administration of IP.
7. Have previously undergone drainage of ascites and/or pleural effusion within 4 weeks prior to screening, or have clinically significant effusions at screening.
8. Have any of the following ocular criteria:

   1. Symptomatic retinal vein occlusion or central serous retinopathy defined as fluid accumulation between the retinal pigment epithelium and the outer segment of the eye
   2. Symptomatic neovascular age related macular degeneration (neovascular/wet age related macular degeneration) or non proliferative diabetic retinopathy with macular edema
   3. Uncontrolled glaucoma, defined as intraocular pressure >21 mmHg despite treatment or history of previous glaucoma filtration surgery
   4. Presence of active intraocular inflammation, uveitis, keratitis, keratoconjunctivitis, keratopathy, corneal abrasion inflammation, or ulceration
   5. Any other clinically significant risk factor for ocular disorders described above
9. Have had major surgery within 4 weeks prior to the first administration of IP. Patients should have recovered from the effects of major surgery or significant traumatic injury within 14 days prior to administration of the IP. Major surgery is defined as requiring more extensive procedure than that including local anesthesia (general anesthesia, respiratory assistance, or regional anesthesia) or open biopsy.
10. Have serious non-healing wounds, ulcers, or bone fractures, except for traumatic fractures not requiring surgical intervention.
11. Have an active infection treated with systemic anti-infectives within 2 weeks prior to the first administration of IP. Prophylactic anti-infectives that are not inhibitors or inducers of CYP3A4 are permitted.
12. Have concurrent unstable or uncontrolled systemic diseases such as the following:

    1. Uncontrolled hypertension despite treatment (systolic blood pressure ≥160 mmHg or diastolic blood pressure ≥100 mmHg)
    2. Clinically significant arrhythmia, unstable angina, congestive heart failure (class III or IV of New York Heart Association), or acute myocardial infarction within 6 months prior to screening
    3. Concurrent active systemic infections requiring systemic antibiotics or antifungals (exception for management of cetuximab-related rash)
    4. Active infections of hepatitis B, hepatitis C, or history of human immunodeficiency virus
    5. Any other chronic disease, which, at the discretion of the investigator, could jeopardize the safety of patients or patients' compliance with the protocol.
    6. Clinically significant venous thromboembolism requiring systemic anticoagulant (exception for prophylactic use)
13. Have a history of gastrointestinal or trachea-esophageal fistulas.
14. Gastrointestinal perforation, non-gastrointestinal fistulas, inflammatory bowel disease, or other bowel diseases accompanying chronic diarrhea within 6 months prior to screening.
15. Current (or planned) pregnancy or breastfeeding from screening to at least 6 months following the last IP administration.
16. Any condition, at the discretion of the investigator, which puts the patient at risk to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-07-14 (Actual); Primary Completion 2025-08-08 (Estimated); Study Completion 2025-08-08 (Estimated)

PRIMARY OUTCOMES:
Incidence of Dose-limiting toxicities (DLT) | During Cycle 1 in Part 1 (each cycle is 28 days)
Incidence of adverse events (AE)/serious adverse events (SAE) | From Baseline to 28 days after last dose

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax) | Cycle 1, Cycle 2, Subsequent Cycles up to 2 years (each cycle is 28 days)
Area under the plasma concentration time curve (AUC) | Cycle 1, Cycle 2, Subsequent Cycles up to 2 years (each cycle is 28 days)
Time to maximum plasma concentration (Tmax) | Cycle 1, Cycle 2, Subsequent Cycles up to 2 years (each cycle is 28 days)
Trough plasma concentration (Ctrough) | Cycle 1, Cycle 2, Subsequent Cycles up to 2 years (each cycle is 28 days)
Elimination half-life (T1/2) | Cycle 1, Cycle 2, Subsequent Cycles up to 2 years (each cycle is 28 days)
Apparent volume of distribution during terminal phase (Vz/F) | Cycle 1, Cycle 2, Subsequent Cycles up to 2 years (each cycle is 28 days)
Accumulation ratio (Rac) | Cycle 1, Cycle 2, Subsequent Cycles up to 2 years (each cycle is 28 days)
Overall response rate (ORR) based on RECIST v1.1 | Screening, Subsequent Cycles (every 8 weeks for 6 month, and then every 12 weeks up to 2 years), within 28 days after last dose (each cycle is 28 days)
Progression-free survival (PFS) | From baseline, every 12 weeks, up to within 28 days after last dose

OTHER OUTCOMES:
Predictive biomarker analyses for genotyping mutation | Screening, Subsequent Cycles up to 2 years, within 28 days after last dose (each cycle is 28 days)

CONTACTS AND LOCATIONS:
Locations (6):
- Australia (3):
  - Monash Medical Center, Clayton, Victoria
  - Austin Hospital, Heidelberg, Victoria
  - Linear Clinical Research Limited, Nedlands, Western Australia
- South Korea (3):
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Severance Hospital, Yonsei University Health System, Seoul
  - Samsung Medical Center, Seoul